CLINICAL TRIAL: NCT00319397
Title: Arterial Stiffness With Age: Part 1 and 2
Brief Title: Effects of Age and Exercise on Blood Pressure Regulation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: J. Andrew Taylor, PhD, Spaulding Rehabilitation Hospital
Other Study IDs: AG0063; R01AG014376 (NIH)
Record Dates: First submitted 2006-04-26; First posted 2006-04-27 (Estimated); Last update posted 2009-12-14 (Estimated); Status verified 2009-01

CONDITIONS: Cardiovascular Disease; Aging
Keywords: vascular resistance; vasomotion; coronary disorder; hemodynamics; physical fitness
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Behavioral: Exercise-Training Program

SUMMARY:
The purpose of this study is to investigate the effects of age, exercise and cardiovascular disease on blood pressure.

DETAILED DESCRIPTION:
This study is being done to find out how age, activity level, and the presence of heart disease affect the way the body controls blood pressure. A total of 80 individuals will be recruited for the study, and will consist of two groups: sedentary healthy individuals and those with coronary artery disease (CAD). Each group will undergo screening tests, including history, questionnaires, physical exam, lab tests, treadmill exercise tolerance test, and maximal exercise test. These screening tests will be repeated at 3 months and 6 months.

The study involves 20 visits over a 6-month period. An exercise-training program will be designed for the individual's fitness level. During the first month, the individual will be supervised while exercising at Spaulding Rehabilitation Hospital, but after that may choose to exercise at home or in a fitness center. These exercise sessions will take place 3-5 times per week for 15-40 minutes per session based on the individual's exercise program, increasing to 4-6 times per week for 30-60 minutes per session after the first month. Participants will be required to visit Spaulding Rehabilitation Hospital a minimum of once every two weeks so that information can be collected from a heart rate monitor.

Testing is done at the beginning and end of the exercise-training intervention period to determine what effect the intervention has had on the individual's blood pressure regulation. This testing consists of 2 sequential study days. During the first day's testing, which will last about 2 hours, the participant will receive 8 low doses of atropine to alter vagal effects. On the second day, which will take about 4 hours, the participant will receive sodium nitroprusside, phenylephrine, and low-dose atropine while sympathetic nervous activity is recorded. Differences in blood pressure regulation pre- and post-training will be studied.

ELIGIBILITY:
Inclusion Criteria:

Sedentary Older Individuals Group:

* Healthy men and women ages 55-75
* Normally physically active (performing regular aerobic exercise less than 60 minutes per week) with aerobic capacities below the 80th percentile for age and gender

Coronary Artery Disease (CAD) Group:

* Men and women ages 55-75
* Written authorization from participant's cardiologist to participate in the study (Note: if Dr. Zervos is the participant's cardiologist, their primary care physician will also be asked to give written authorization)
* Documented CAD by previous MI or angiography

Exclusion Criteria:

General exclusion criteria for all groups:

* Neurological diseases
* Diabetes
* History of migraine headaches
* Hypertension
* Glaucoma
* Pacemaker
* History of stroke or TIA
* High cholesterol
* Current cancer
* Benign prostatic hyperplasia
* Allergy to sulfa
* Carotid disease
* Currently taking anti-depression, anti-psychotic, or anti-anxiety medications

Sedentary Older Individuals Group:

* Coronary artery or carotid vascular disease

Coronary Artery Disease (CAD) Group:

* Myocardial Infarction (MI), Percutaneous Transluminal Coronary Angioplasty (PTCA) or Coronary Artery Bypass Graft (CABG) in the last 3 months
* Unstable angina, EF branch block severe valvular disease, chronic atrial fibrillation, and frequent atrial or ventricular arrhythmias (including more than 3 PVCs or APCs per minute)
* Currently taking anticoagulants or any cardioactive medications other than ACE inhibitors, calcium channel blockers, and beta-blockers

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2004-04; Study Completion 2007-03

CONTACTS AND LOCATIONS:
Overall Officials: J. Andrew Taylor, PhD, Principal Investigator — Spaulding Rehabilitation Hospital, Harvard Medical School; Gerasimos Zervos, MD, Principal Investigator — Chief of Nuclear Cardiology, Massachusetts General Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Hagbarth KE, Vallbo AB. Pulse and respiratory grouping of sympathetic impulses in human muscle-nerves. Acta Physiol Scand. 1968 Sep-Oct;74(1):96-108. doi: 10.1111/j.1748-1716.1968.tb04218.x. No abstract available. PMID 4235387
- [Background] Wallin BG, Fagius J. Peripheral sympathetic neural activity in conscious humans. Annu Rev Physiol. 1988;50:565-76. doi: 10.1146/annurev.ph.50.030188.003025. No abstract available. PMID 3288106
- [Background] Eckberg DL, Wallin BG, Fagius J, Lundberg L, Torebjork HE. Prospective study of symptoms after human microneurography. Acta Physiol Scand. 1989 Dec;137(4):567-9. doi: 10.1111/j.1748-1716.1989.tb08804.x. No abstract available. PMID 2690582
- [Background] Yuasa T, Takata S, Maruyama M, Yasuma K, Yoshizawa H, Kontani M, Nagai H, Sakagami S, Kobayashi K. Low-dose atropine attenuates muscle sympathetic nerve activity in healthy humans. Hypertens Res. 2000 May;23(3):213-8. doi: 10.1291/hypres.23.213. PMID 10821129
- [Background] Ikuta Y, Shimoda O, Kano T. Quantitative assessment of the autonomic nervous system activities during atropine-induced bradycardia by heart rate spectral analysis. J Auton Nerv Syst. 1995 Mar 18;52(1):71-6. doi: 10.1016/0165-1838(94)00148-d. PMID 7782571
- [Background] Alcalay M, Izraeli S, Wallach-Kapon R, Tochner Z, Benjamini Y, Akselrod S. Paradoxical pharmacodynamic effect of atropine on parasympathetic control: a study by spectral analysis of heart rate fluctuations. Clin Pharmacol Ther. 1992 Nov;52(5):518-27. doi: 10.1038/clpt.1992.180. PMID 1424426
- [Background] Smyth HS, Sleight P, Pickering GW. Reflex regulation of arterial pressure during sleep in man. A quantitative method of assessing baroreflex sensitivity. Circ Res. 1969 Jan;24(1):109-21. doi: 10.1161/01.res.24.1.109. No abstract available. PMID 4303309